CLINICAL TRIAL: NCT03932240
Title: In Vivo Effects of Fibrinogen Concentrate (FC) Versus Cryoprecipitate on the Neonatal Fibrin Network Structure After Cardiopulmonary Bypass (CPB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Laura A Downey, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00109310
Record Dates: First submitted 2019-04-03; First posted 2019-04-30 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Hemostasis
Keywords: Fibrinogen Concentrate; FC; Cryoprecipitate; Transfusion; in vivo; Open-heart surgery; Cardiopulmonary Bypass; Fibrin Network Structure
MeSH Terms: interventions — Fibrinogen; cryoprecipitate coagulum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fibrinogen Concentrate (FC) (Experimental): Neonates undergoing elective cardiac surgery requiring cardiopulmonary bypass (CPB) who are randomized to receive platelets and FC after separation from bypass. The dose of fibrinogen concentrate will be calculated to achieve a level of 300mg/dL after drug administration.
  If a patient in either arm continues to have post-bypass bleeding, the anesthesiologist will use point of care testing and the transfusion thresholds outlines in the transfusion algorithm to determine appropriate products for transfusion.
  Interventions: Drug: Fibrinogen Concentrate (FC)
- Cryoprecipitate (Active Comparator): Neonates undergoing elective cardiac surgery requiring cardiopulmonary bypass (CPB) who are randomized to receive platelets and cryoprecipitate. Standard transfusion algorithm includes two units of cryoprecipitate, which result in a median post-operative fibrinogen level of 286mg/dL (based on findings by Downey et al., published in Anesthesia and Analgesia in 2020).
  If a patient in either arm continues to have post-bypass bleeding, the anesthesiologist will use point of care testing and the transfusion thresholds outlines in the transfusion algorithm to determine appropriate products for transfusion.
  Interventions: Drug: Cryoprecipitate

INTERVENTIONS:
Drug: Fibrinogen Concentrate (FC) — The dose of fibrinogen concentrate will be calculated to achieve a level of 300mg/dL after drug administration.
  Other Names: RiaSTAP
  Arms: Fibrinogen Concentrate (FC)
Drug: Cryoprecipitate — The standard transfusion algorithm includes two units of cryoprecipitate, which result in a median post-operative fibrinogen level of 286mg/dL.
  Arms: Cryoprecipitate

SUMMARY:
This primary aim of this study is to compare the in vivo effects of fibrinogen concentrate and cryoprecipitate on the neonatal fibrin network after surgery with cardiopulmonary bypass to develop effective and safe strategies for managing coagulopathies in neonates.

DETAILED DESCRIPTION:
This study is a prospective, randomized control trial comparing two different sources of fibrinogen on clot kinetics (degradation and structure) in post-CPB coagulopathy in neonates undergoing cardiac surgery. The two sources of fibrinogen include the blood product, cryoprecipitate, and a blood product alternative, fibrinogen concentrate. Cryoprecipitate is an allogenic blood product that requires cross-matching and thawing prior to administration and is associated with immunologic reactions and possible pathogen transmission. Fibrinogen concentrate, a blood product alternative, is a purified form of fibrinogen, which undergoes a pasteurization process to minimize the risk of immunologic and allergic reactions. The primary aim of this study is compare the in vivo effect of post-CPB administration of FC, a blood product alternative, to cryoprecipitate on neonatal clot properties and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Full term neonates (36-42 weeks gestational age)
2. Infants =< 30 days of age at time of surgery
3. APGAR score of 6 or greater at 5 minutes after delivery
4. Neonates undergoing elective cardiac surgery requiring CPB at Children's Healthcare of Atlanta
5. Parents willing to participate and able to understand and sign the provided informed consent

Exclusion Criteria:

1. Preterm neonates (less than 36 weeks gestation)
2. Patients undergoing an emergent procedure or surgery not requiring CPB
3. Patients with personal or family history of a coagulation defect or coagulopathy
4. Parents unwilling to participate or unable to understand and sign the provided informed consent

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Downey, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta (CHOA), Egleston, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices), will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved protocol. Proposals should be directed to laura.ansley.downey@emory.edu. To gain access, data requestors will need to sign and obtain a data use agreement. The data will be available for five years in the investigator's Emory's data warehouse.

REFERENCES:
- [Derived] Downey LA, Moiseiwitsch N, Nellenbach K, Xiang Y, Brown AC, Guzzetta NA. Effect of In Vivo Administration of Fibrinogen Concentrate Versus Cryoprecipitate on Ex Vivo Clot Degradation in Neonates Undergoing Cardiac Surgery. Anesth Analg. 2025 Aug 1;141(2):240-251. doi: 10.1213/ANE.0000000000007123. Epub 2024 Aug 8. PMID 39116012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta (CHOA) at Egleston in Atlanta, Georgia, USA. Participant enrollment began August 13, 2019 and all follow up was complete by November 16, 2021.
Groups:
- Fibrinogen Concentrate (FC): Neonates undergoing elective cardiac surgery requiring cardiopulmonary bypass (CPB) who were randomized to receive platelets and fibrinogen concentrate after separation from bypass.
- Cryoprecipitate: Neonates undergoing elective cardiac surgery requiring cardiopulmonary bypass (CPB) who were randomized to receive platelets and cryoprecipitate after separation from bypass.
Period: Overall Study
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Started | 18 | 18
Completed Study Per Protocol | 17 | 13
Completed (Intent to Treat Population) | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 18 | 36
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 9 | 14 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36
Weight [Median (Inter-Quartile Range); unit: kilograms (kg)] | 3.10 [2.66 to 3.58] | 3.50 [2.92 to 3.69] | 3.40 [2.68 to 3.69]

OUTCOME MEASURES:

1. Primary Outcome: Clot Degradation at 24 Hours Post-operatively
Description: Blood samples were obtained from an arterial line that was required for the planned surgical procedure. Samples were centrifuged to yield platelet poor plasma (PPP), stored at -80 degrees Celsius and utilized for the clot analysis. Clot degradation was determined by degradation kinetic study. Blood samples were collected at four time points:1) baseline sample within 24 hours of surgery and after induction of anesthesia prior to CPB; 2) after termination of CPB and transfusion of platelets and either cryoprecipitate or fibrinogen (within 1 hour of separation from bypass; 3) upon arrival to the ICU; 4) 24 hours post-operatively. The primary outcome is to examine differences in clot degradation between study arms at 24 hours post-surgery.
Time Frame: From induction of anesthesia to 24 hours postoperatively
Population: This analysis includes the Intent to Treat Population, which is comprised on all participants regardless of if they completed the study per protocol.
Measure: Median (Inter-Quartile Range); unit: microns per hour
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
microns per hour
  After induction of anesthesia prior to CPB | 0.65 [0.41 to 1.49] | 0.88 [0.37 to 1.42]
  After termination of CPB and transfusion of platelets and either cryoprecipitate or fibrinogen | 0.78 [0.33 to 0.92] | 0.46 [0.27 to 1.56]
  Upon arrival to the ICU | 0.65 [0.44 to 0.88] | 0.55 [0.28 to 2.39]
  24 hours post-operatively | 0.92 [0.55 to 1.42] | 0.76 [0.34 to 1.22]

2. Secondary Outcome: Clot Strength
Description: Blood samples will be obtained from an arterial line that is required for the planned surgical procedure. They will be centrifuged to yield platelet poor plasma (PPP), stored at -80 degrees Celsius and utilized for the clot analysis. Strength will be assessed by rheology and atomic force microscopy (AFM).
Time Frame: From induction of anesthesia to 24 hours postoperatively
Population: Unfortunately, due to the required amount of blood necessary for triplicates of the primary outcome, there was not enough blood to examine clot strength. Due to the small amount of blood collected from neonates the samples were used for the outcome measures with the highest priority and the amount of remaining blood was not sufficient to assess clot strength.
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Clot Polymerization Kinetic
Description: Blood samples will be obtained from an arterial line that is required for the planned surgical procedure. They will be centrifuged to yield platelet poor plasma (PPP), stored at -80 degrees Celsius and utilized for the clot analysis. Polymerization will be determined by thrombin-initiated turbidity/absorbency curves.
Time Frame: From induction of anesthesia to 24 hours postoperatively
Population: Due to the maximum allowable blood to be taken from a neonate, there was not enough remaining blood available to examine clot polymerization kinetics. In order to carry out the degradation assay on neonatal fibrinogen, the study team improved the assay they originally intended to use and no longer did polymerization assays as part of the degradation assay. Due to the change in the degradation assay, the team was not able to collect additional blood for the clot polymerization kinetics assay.
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Fibrin Fiber Alignment
Description: Clot structure is assessed by examination of images of clot fibrin fiber alignment. Quantification of clot fiber alignment was achieved through the application of an automated algorithm based on a fast Fourier transform that measures the alignment of the fibers, as well as visual inspection. A reference range has not been established for neonates, however, higher values indicate more dense clot structure.
Time Frame: From induction of anesthesia to 24 hours postoperatively
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: black/white pixels
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
black/white pixels
  After induction of anesthesia prior to CPB | 0.46 [0.26 to 0.61] | 0.54 [0.32 to 0.68]
  After termination of CPB and transfusion of platelets and either cryoprecipitate or fibrinogen | 0.52 [0.37 to 0.59] | 0.54 [0.45 to 0.63]
  Upon arrival to the ICU | 0.41 [0.31 to 0.58] | 0.44 [0.37 to 0.66]
  24 hours post-operatively | 0.37 [0.15 to 0.52] | 0.38 [0.10 to 0.58]

5. Secondary Outcome: Interoperative Transfusion Requirement
Description: Blood product transfusion requirements were obtained from electronic medical records. An increased transfusion requirement indicates increased interoperative bleeding, thus, lower values are preferable.
Time Frame: During surgery (up to 6 hours)
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
ml/kg | 27.2 [19.0 to 36.9] | 41.6 [29.2 to 52.4]

6. Secondary Outcome: Transfusion Requirements Within the First 24 Hours After Surgery
Description: Transfusion requirements within the first 24 hours of surgery were obtained from electronic medical records.
Time Frame: 24 hours postoperatively
Population: The recording of transfusions in the intensive care unit (ICU) changed in the middle of this study and therefore transfusions were not consistently documented by the clinical staff, thus, the study investigators decided to not collect information about transfusions up to 24 hours after surgery from medical records as data could not be reliably analyzed.
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Amount of Post-operative Bleeding
Description: Post-operative bleeding was recorded by 24 hour chest tube output. Higher values indicate greater post-operative bleeding.
Time Frame: Up to 24 hours postoperatively
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
ml/kg | 38.5 [32.0 to 70.5] | 45.5 [31.5 to 69.0]

8. Secondary Outcome: Mechanical Ventilation Time
Description: Mechanical ventilation time was obtained from medical records. Higher values indicate increased need for mechanical ventilation.
Time Frame: Time of extubation (up to 2 weeks)
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
hours | 63.3 [35.6 to 77.9] | 117.2 [39.9 to 168.0]

9. Secondary Outcome: Length of ICU Stay
Description: Length of ICU stay was obtained from medical records. A shorter ICU stay indicates a favorable state of health.
Time Frame: At discharge from ICU (typically up to 21 days)
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
days | 7.0 [5.0 to 14.0] | 8.5 [5.3 to 13.3]

10. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay was obtained from medical records. A shorter hospital stay indicates a favorable state of health.
Time Frame: At discharge from hospital (up to 150 days)
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
days | 16.0 [10.8 to 47.5] | 14.5 [9.5 to 29.8]

11. Secondary Outcome: Number of Adverse Events
Description: Adverse events within seven days of surgery were obtained from medical records.
Time Frame: Within seven days of surgery
Population: This analysis includes the Intent to Treat Population.
Measure: Number; unit: adverse events
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
adverse events | 6 | 11

12. Other Pre Specified Outcome: Number of Events of Postoperative Thrombosis
Description: The number of events of clinically significant postoperative thrombosis that required treatment were obtained from medical records.
Time Frame: Within the first 24 hours of surgery
Population: This analysis includes the Intent to Treat Population.
Measure: Number; unit: events
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
events | 2 | 2

13. Other Pre Specified Outcome: Fibrinogen Plasma Level
Description: Blood samples were obtained from an arterial line that was required for the planned surgical procedure. The samples were centrifuged to yield platelet poor plasma (PPP), stored at -80 degrees Celsius and utilized for the clot analysis. ELISA was used to measure coagulation factors at each time point. Normal fibrinogen plasma values are between 0.5 to 15 mcg/mL.
Time Frame: From induction of anesthesia to 24 hours postoperatively
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
mcg/mL
  Within 2 hours of induction of anesthesia prior to CPB | 1.39 [0.99 to 2.11] | 1.09 [0.75 to 2.20]
  After termination of CPB and transfusion of platelets and either cryoprecipitate or fibrinogen | 1.26 [0.99 to 1.57] | 1.97 [1.12 to 2.82]
  Upon arrival to the ICU | 1.42 [1.08 to 2.22] | 1.28 [1.07 to 1.69]
  24 hours post-operatively | 1.76 [1.49 to 2.11] | 1.87 [1.43 to 2.27]

14. Other Pre Specified Outcome: Thrombin Plasma Level
Description: Blood samples were obtained from an arterial line that was required for the planned surgical procedure. The samples were centrifuged to yield platelet poor plasma (PPP), stored at -80 degrees Celsius and utilized for the clot analysis. ELISA was used to measure coagulation factors at each time point. The reference range for thrombin plasma level is 0.000313 to 0.02 mcg/mL.
Time Frame: From induction of anesthesia to 24 hours postoperatively
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
mcg/mL
  Within 2 hours of induction of anesthesia prior to CPB | 0.02 [0.01 to 0.06] | 0.07 [0.02 to 0.10]
  After termination of CPB and transfusion of platelets and either cryoprecipitate or fibrinogen | 0.02 [0.01 to 0.05] | 0.05 [0.03 to 0.06]
  Upon arrival to the ICU | 0.03 [0.02 to 0.06] | 0.05 [0.03 to 0.06]
  24 hours post-operatively | 0.02 [0.01 to 0.08] | 0.06 [0.03 to 0.08]

15. Other Pre Specified Outcome: FXIII Plasma Level
Description: Blood samples were obtained from an arterial line that was required for the planned surgical procedure. The samples were centrifuged to yield platelet poor plasma (PPP), stored at -80 degrees Celsius and utilized for the clot analysis. ELISA was used to measure coagulation factors at each time point. The reference range for FXIII plasma level is 0.000469 to 0.03 mcg/mL.
Time Frame: From induction of anesthesia to 24 hours postoperatively
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
mcg/mL
  Within 2 hours of induction of anesthesia prior to CPB | 0.03 [0.03 to 0.06] | 0.03 [0.03 to 0.04]
  After termination of CPB and transfusion of platelets and either cryoprecipitate or fibrinogen | 0.04 [0.02 to 0.05] | 0.04 [0.03 to 0.07]
  Upon arrival to the ICU | 0.04 [0.03 to 0.06] | 0.05 [0.04 to 0.07]
  24 hours post-operatively | 0.03 [0.03 to 0.04] | 0.04 [0.03 to 0.05]

16. Other Pre Specified Outcome: Von Willebrand Factor Plasma Level
Description: Blood samples were obtained from an arterial line that was required for the planned surgical procedure. The samples were centrifuged to yield platelet poor plasma (PPP), stored at -80 degrees Celsius and utilized for the clot analysis. ELISA was used to measure coagulation factors at each time point. Lower values may indicate an increased risk of excessive bleeding.
Time Frame: From induction of anesthesia to 24 hours postoperatively
Population: This analysis includes the Intent to Treat Population.
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
Number analyzed (Participants) | 18 | 18
IU/mL
  Within 2 hours of induction of anesthesia prior to CPB | 2.98 [1.86 to 7.01] | 4.68 [1.75 to 6.56]
  After termination of CPB and transfusion of platelets and either cryoprecipitate or fibrinogen | 4.43 [3.48 to 15.56] | 6.11 [5.42 to 16.37]
  Upon arrival to the ICU | 5.06 [3.43 to 7.16] | 6.15 [5.53 to 12.81]
  24 hours post-operatively | 3.95 [3.35 to 12.75] | 7.00 [4.78 to 11.73]

ADVERSE EVENTS:
Time Frame: Information on serious and non-serious adverse events was collected beginning at the time consent to participate in the study was given through 7 days post-surgery. Mortality was collected until the participant was discharged from the hospital (up to 150 days).
Arm/Group | Fibrinogen Concentrate (FC) | Cryoprecipitate
All-Cause Mortality (participants affected / at risk) | 1/18 | 1/18
Serious Adverse Events (participants affected / at risk) | 2/18 | 9/18
Other Adverse Events (participants affected / at risk) | 4/18 | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrinogen Concentrate (FC) (N=18) | Cryoprecipitate (N=18)
Extracorporeal membrane oxygenation (ECMO) within 24 hours (Surgical and medical procedures) | 0 | 4
Tamponade (Surgical and medical procedures) | 0 | 1
Chest exploration (Surgical and medical procedures) | 1 | 2
Stroke (Vascular disorders) | 1 | 0
Infection (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrinogen Concentrate (FC) (N=18) | Cryoprecipitate (N=18)
Arrhythmia (Cardiac disorders) | 2 | 4
Thrombosis (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT03932240/Prot_001.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT03932240/SAP_002.pdf